CLINICAL TRIAL: NCT01978652
Title: A Two-Arm, Open-Label, Single-Dose, Phase 1 Study of the Pharmacokinetics, Safety, and Tolerability of Peginterferon Beta-1a (BIIB017) in Japanese and Caucasian Adult Healthy Subjects
Brief Title: Pharmacokinetic Study of Peginterferon Beta-1a in Japanese and Caucasian Adult Healthy Participants.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 105HV104; 2013-002912-28
Record Dates: First submitted 2013-11-01; First posted 2013-11-07 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Healthy
MeSH Terms: interventions — peginterferon beta-1a

ARMS (2):
- Peginterferon Beta-1a administered to Japanese participants (Experimental): A single dose of Peginterferon Beta-1a 125 μg subcutaneous (SC) injection administered by pre-filled syringe
  Interventions: Biological: Peginterferon Beta-1a
- Peginterferon Beta-1a administered to Caucasian participants (Experimental): A single dose of Peginterferon Beta-1a 125 μg subcutaneous (SC) injection administered by pre-filled syringe
  Interventions: Biological: Peginterferon Beta-1a

INTERVENTIONS:
Biological: Peginterferon Beta-1a — As specified in the treatment arm
  Other Names: Plegridy; BIIB017

SUMMARY:
The primary objective of this study is to characterise the pharmacokinetics (PK) of BIIB017 (Peginterferon Beta-1a) administered as a single 125 μg subcutaneous (SC) dose in Japanese and Caucasian adult healthy participants. The secondary Objective is to assess the safety and tolerability of a single 125 μg subcutaneous (SC) dose of BIIB017 in Japanese and Caucasian adult healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a BMI of 19 to 29 kg/m2, inclusive, and minimum body weight of 45.0 kg at Screening and at Baseline.
* Japanese subjects must have been born in Japan and have both parents and grandparents of Japanese origin. Additionally, Japanese subjects should have lived outside of Japan for less than 5 years and maintained a similar diet since leaving Japan (to be verified by a questionnaire at Screening).
* Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 90 days after their last dose of study treatment.
* Non smoker or be willing to abstain from using tobacco and tobacco-containing products for 24 hours prior to clinic admission and during the In-Clinic Period and to smoke no more than 10 cigarettes (or equivalent) per day throughout the remainder of the study.
* Must be willing to refrain from all alcohol consumption for 48 hours prior to Day 1 and during the In-Clinic Period and to limit the intake of alcohol to no more than 2 units per day throughout the remainder of the study.

Key Exclusion Criteria:

* Known history of, or positive test result at Screening for human immunodeficiency virus (HIV).
* Known history of, or positive test result for hepatitis C virus (test for hepatitis C virus antibody [HCV Ab]) or hepatitis B virus (test for hepatitis B surface antigen [HBsAg]).
* Subjects with a history of malignant disease, including solid tumours and haematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured or subjects with cervical cancer stage 0 if completely excised).
* History of severe allergic or anaphylactic reactions in the opinion of the Investigator.
* Known allergy to any interferon or any component of BIIB017.
* History of suicidal ideation or an episode of clinically significant depression (as determined by the Investigator) within 3 months prior to Day 1.
* Any previous treatment with prescription or investigational pegylated drugs. The prior use of over-the-counter pegylated products, including cosmetics, is allowed.
* Previous treatment with any interferon product.
* History of hypersensitivity or intolerance to paracetamol, ibuprofen, or naproxen, that would preclude use of at least 1 of these during the study.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2013-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity (AUC0-∞) | Up to 240 hours post-dose

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of Peginterferon Beta-1a | Up to 240 hours post-dose
Number of participants that experience adverse events (AEs) and serious adverse events (SAEs) | Up to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Leeds, West Yorkshire, United Kingdom